CLINICAL TRIAL: NCT05870293
Title: THE EFFECT OF GOAL-SETTING DIABETES NURSE COACHING ON HbA1c VALUE AND STRENGTHENING DIABETES
Brief Title: EFFECT OF DIABETES NURSE COACHING ON DIABETES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuğba Bilgehan (Other)
Responsible Party: Sponsor-Investigator, Tuğba Bilgehan, Asst Prof, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TUGBABILGEHAN2
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Nurse's Role; Diabetes Mellitus, Type 2
Keywords: walt disney; nurse coaching; nursing
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESPONSE GROUP (Experimental): The study will be done online and the application will be explained to the patients. Randomly selected groups will be made using a single-blind technique, not knowing which group is the intervention group. Pre-test will be applied to the diabetic patients included in the experimental groups and control groups. After the preliminary tests are applied to the individuals with diabetes in the intervention 1 group, a nurse coaching interview will be held with diabetes by applying the 'walt disney' method. In accordance with the principles of coaching, 2 sessions will be held under the management of the patient. After the first session, 10 days later, in the second session, life coaching with diabetes will be done with the Walt Disney method. After 10 days after the 2nd interview, the final tests will be applied at the end of the 1st month.
  Interventions: Behavioral: nurse coaching
- control group (No Intervention): The control group will be given a pre-test and a post-test 1 month later without any intervention.

INTERVENTIONS:
Behavioral: nurse coaching — 2 sessions of nurse coaching including the Walt Disney method will be applied to the participants.
  Arms: RESPONSE GROUP

SUMMARY:
American Diabetes Association and American Clinical Endocrinology American Association of Clinical Endocrinologists, treatment and care of individuals with diabetes in achieving their goals; regulation of nutrition, regulation of physical activity, pharmacological treatment, diabetes education, continuous monitoring and health checks should be done.

emphasizes (3,4). Individuals with diabetes receive diabetes self-management education and support when necessary.

they should. Diabetes self-management is the knowledge, skills and abilities necessary for the individual's self-care.

It is defined as the facilitation process (4,5). Competent and skilled in self-management individuals with diabetes can improve their health outcomes. American Diabetes Association (ADA), diabetes self-management education necessary for the self-care of people with diabetes.

take an individual-centered approach and make joint decisions to facilitate knowledge, skills and abilities It defines it as a process based on diagnosis, starting at the diagnosis stage and continuing (5).

The goal of diabetes self-management is to introduce new skills and abilities that support diabetes patients' self-management goals.

Developing behaviors and forming habits. General objectives of diabetes self-management education On the other hand, it enables individuals diagnosed with diabetes to make informed decisions, problem solving, personal care behavior, metabolic outcomes, health status and quality of life to improve (5). To strengthen the diabetes patient by providing self-management needs knowledge, skills and motivation about the disease. Counseling for nurses ability of the patient to adapt to his/her illness and self-care by doing and educating provides access (6). Coaching sessions to strengthen diabetes self-management and diabetes is applied. The coach is committed to maximizing the client's strengths, To ensure that it is used fully through continuous education, to be more effective, new to develop skills and activities, to be ready for new responsibilities, and to self-management.

It is the person who provides the necessary motivation (7). Life Coaching with Diabetes, about lifestyle with diabetes professional life coaching practices, aiming at behavior change in approaches (ICF-International Coaching Federation) is based on the basic principles and principles. life with diabetes coaching is used to help people who have been diagnosed with diabetes make the necessary changes in life through coaching.

to give practical applications. Walt Disney is a goal setting coaching exercise. The work consists of 6 steps. These steps it is as follows.

1. Detection of the subject and 3 anchor methods
2. Dreamer + Ground Anchor + Separator
3. Planner + Ground Anchor + Separator
4. Critic + Ground Anchor + Separator
5. Brainstorming
6. Metatest

DETAILED DESCRIPTION:
Expected benefits:

Diabetes is a non-communicable disease that is increasing rapidly day by day. Providing support integrated with life coaching with diabetes will increase the awareness of people with diabetes and enable them to manage their diabetes.

* Developing appropriate self-care activities (physical activity, medical nutrition, drug management, avoiding risky behaviors, etc.) by improving the self-management skills of the individual with diabetes,
* The individual with diabetes becomes self-managing self-care practices,
* Improving decision-making and problem-solving skills of individuals with diabetes,

H0: Diabetes nurse coaching given to individuals with Type 2 Diabetes has no effect on HbA1c value and on strengthening diabetes.

H1: Diabetes nurse coaching given to individuals with Type 2 Diabetes has an effect on HbA1c value and strengthening diabetes.

The Universe of the Research The population of the study consists of patients with Type 2 Diabetes between the ages of 18-64 who applied to Ankara Pursaklar State Hospital Internal Medicine outpatient clinic.

Sample Selection of the Research The sample size was calculated using G*Power Software (ver. 3.1.9.7). The effect size was calculated by using the mean and standard deviation values of the last test of the experimental and control groups of the 'Diabetes strengthening scale' used in the randomized controlled study by Zamanzadeh (2017), the sample of the study. The sample size required for the study was calculated as 34 patients, 17 patients for each group, in the power analysis performed with 95% confidence level and 5% tolerance. However, it was aimed to reach 21 individuals from each group with the foresight that there may be participant losses during the study process. To avoid bias in assigning the individuals to be included in the study to the groups, https://randomizer.org/ With the help of the help of 1-42, random numbers were generated as 2 groups and the incoming individuals will be assigned to the relevant groups.

Data Collection Technique and Tools The data in the research will be collected through the data collection form, the diabetes empowerment scale, which was prepared based on the researcher's experiences and the literature.

1. Data collection form: It will be created by the researcher based on the literature. (such as age, gender, how many years have had diabetes).
2. Diabetes empowerment scale: The scale developed by Özcan and Korkmaz (2012); It has 3 sub-dimensions: management of psychosocial aspects in diabetes, level of dissatisfaction and readiness for change, setting and achieving diabetes goals.

ELIGIBILITY:
Inclusion Criteria:

* Who voluntarily agrees to participate in the study,

  * Having a smart phone and using it actively,
  * Those between the ages of 18-65,
  * The patient who was diagnosed with type 2 diabetes at least 1 year ago,
  * The individual with type 2 diabetes has not developed any chronic complications,
  * HbA1c > 6.5
  * Absence of any psychiatric problems.

Exclusion Criteria:

* not attending the coaching interview
* unwillingness to quit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Diabetes potentiation scale | 1 month
  It consists of 3 sub-dimensions including management of psychosocial aspects in diabetes, level of dissatisfaction and readiness for change, determination and achievement of diabetes goals, and 28 items in total. The highest possible score is 140 and the lowest score is 28. A high score from the scale indicates the strength of diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Bilgehan, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No